CLINICAL TRIAL: NCT06806306
Title: Assessment of the Preoperative Risk Factors for the Development of Post-LASIK Ectasia
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Walid Shaban Abdella, Prinicipal Investigator, Al-Azhar University
Other Study IDs: Post-LASIK Ectasia
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Lasik Eye Surgery
MeSH Terms: interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: LASIK — Laser-assisted in situ keratomileusis is one of the most widely performed refractive surgeries for correcting myopia, hyperopia, and astigmatism

SUMMARY:
: Laser-assisted in situ keratomileusis (LASIK) is one of the most widely performed refractive surgeries, offering effective and long-lasting correction for visual refractive errors. While LASIK has a high success rate and is generally safe, post-LASIK ectasia remains a rare but serious complication that compromises visual outcomes. Several risk factors for post-LASIK ectasia have been identified. The aim of the present study is to determine the preoperative risk factors for the development of post-LASIK ectasia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of corneal ectasia was made by progressive central or inferior corneal steepening, increased myopia and/or astigmatism, and decreased visual acuity

Exclusion Criteria:

* Subjects who had glaucoma diagnosis, other corneal surgeries (other than LASIK), and central corneal opacity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: LASIK patients
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Randleman ectasia score | At the baseline